CLINICAL TRIAL: NCT05416008
Title: A Prospective Observational Study on the Relationship Between Long-term Oral Anti Hepatitis B Nucleoside Analogs and Hepatic Steatosis
Brief Title: The Relationship Between Long-term Oral Anti Hepatitis B Nucleoside Analogs and Hepatic Steatosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Zhangdz2021
Record Dates: First submitted 2022-05-23; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: treatment with ETV: The patients in this group were composed of patients with chronic hepatitis B who firstly take entecavir for the treatment of chronic hepatitis B.
  Take Entecavir capsule orally for a long time, once a day, 0.5mg each time.
- Group 2: treatment with TAF: The patients in this group were composed of patients with chronic hepatitis B who firstly take Tenofovir alafenamide Fumarate for the treatment of chronic hepatitis B.
  Take Tenofovir alafenamide Fumarate tablets orally for a long time, 25mg once a day.
- Group 3: treatment with TDF: The patients in this group were composed of patients with chronic hepatitis B who firstly take Tenofovir disoproxil Fumarate for the treatment of chronic hepatitis B.
  Tenofovir disoproxil fumarate was orally administered for a long time, once a day, 300mg each time.

SUMMARY:
This study aims to investigate whether long-term use of nucleotide analogues could promote hepatic steatosis in patients with chronic hepatitis B. The degree of hepatic steatosis was observed after 3 years of antiviral treatment with nucleoside (acid) analogues for the first time to determine whether the long-term use of anti hepatitis B nucleoside (acid) analogues could promote hepatic steatosis. To explore the anti hepatitis B nucleotide analogues that can promote liver steatosis, so as to provide evidence-based medical evidence for the selection or adjustment of anti hepatitis B virus drugs in patients with chronic hepatitis B.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational study involving chronic hepatitis B patients from the Second Affiliated Hospital of Chongqing Medical University.

Research implementation process and route

Recruitment object: Patients with chronic hepatitis B, defined as persistent hepatitis B surface antigen positive for ≥ 6 months, (aged ≥ 18, treatment-naive ) were consecutively recruited for outpatient routine examination between July 2021 and December 2022. We excluded patients with prior history of hepatocellular carcinoma, concomitant hepatitis C virus or human immunodeficiency virus infection, primary biliary cirrhosis, Wilson's disease, autoimmune hepatitis, significant alcohol intake (≥ 30 g per day for male, or ≥ 20 g per day for female), on steatogenic medications, prior liver transplantation. The basic information and various examination indexes of the patients were collected, and the patients were informed that they needed to go to the outpatient clinic of our hospital for follow-up examination every 1 year, with a total follow-up of 3 years.

Data to be collected: general medical history characteristics: medical record number, name, gender, age, , enrollment time, contact information, and name of anti hepatitis B drugs. Examination and inspection indicators: liver function, renal function, blood chart analysis, blood lipid, hepatitis B two half and half, anti hepatitis C virus, anti hepatitis D virus, AIDS syphilis screening, high precision hepatitis B virus-DNA quantification, abdominal color Doppler ultrasound (if necessary CT or MR), transient elastography of the liver.

Follow up: after enrollment, the relevant examination indexes were rechecked every 1 year. The follow-up period was 3 years.

Statistical analysis: after a three-year follow-up, the data collected were tested by t-test and multivariate Cox analysis to analyze whether the long-term use of anti hepatitis B nucleoside (acid) analogues could promote hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent.
* Male or female.
* 18 ≤ age≤ 80.
* Clinical diagnosis of chronic hepatitis B.
* Has not received anti HBV treatment.

Exclusion Criteria:

* With prior history of HCC
* Concomitant HCV or HIV
* Primary biliary cholangitis
* Wilson's disease
* Autoimmune hepatitis
* Significant alcohol intake (≥ 30 g per day for male, or ≥ 20 g per day for female)
* Taking steatogenic medications
* Prior liver transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis B patients who meet the inclusion conditions and don't meet the exclusion conditions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal color Doppler ultrasound (if necessary CT or MR) | once a year up to 3 years
  Patients with fatty liver were evaluated by abdominal color Doppler ultrasound
Liver transient elastography | once a year up to 3 years
  The CAP value was obtained from the liver transient elastography. According to the CAP value, steatosis is divided into mild (CAP 248-267 dB / m), moderate (CAP 268-279 dB / m) and severe (≥ 280 dB / m).
Lipid profiles | once a year up to 3 years
  Lipid profiles, such as total cholesterol (TC), triglycerides(TG), high-density lipoprotein cholesterol(HDL-C), and low-density lipoprotein cholesterol(LDL-C).

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Zhang, Doctor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no sharing plan